CLINICAL TRIAL: NCT05515770
Title: An Implementation Study of Long-acting Injectable Cabotegravir (CAB-LA) for HIV Pre-Exposure Prophylaxis (PrEP) Among Young MSM, Non-binary and Transgender Persons (The ImPrEP CAB Study)
Brief Title: The Implementation of Pre-exposure Prophylaxis of Injectable Cabotegravir
Acronym: ImPrepCab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Evandro Chagas National Institute of Infectious Disease (Other)
Collaborators: Beatriz Grinsztejn (Unknown); Thiago Torres (Unknown); Valdilea Gonçalves (Unknown); Brenda Hoagland (Unknown)
Responsible Party: Principal Investigator, Raquel Malaguthi de Souza, Beatriz Grinsztejn, MD, PhD, Evandro Chagas National Institute of Infectious Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 59166522.7.1001.5262
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: Cabotegravir; pre exposure prophylaxis
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Intervention Model Description: We will use both quantitative (surveys, laboratory tests, service statistics) and qualitative (in-depth interviews and focus group discussions) methods. HIV incidence in the CAB LA cohort (N=1200) in this study will be compared with a similar cohort accessing oral PrEP through the public health system. The effectiveness of the mHealth intervention will be assessed using interrupted time series analysis. The WhatsApp intervention will be randomized at the individual level and data analyzed using logistic mixed models.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Injectable Cabitegravir (Experimental): Participants that are interested in Cab long action injectable
  Interventions: Drug: Cabotegravir Injection

INTERVENTIONS:
Drug: Cabotegravir Injection — Long action cabotegravir injection
  Other Names: brand name: Apretude

SUMMARY:
Although CAB LA PrEP has been proven efficacious in blinded randomized controlled clinical trials, additional research is needed to evaluate effectiveness in real world settings as well as to identify effective implementation strategies. The proposed implementation study will assess the safety and effectiveness of open label CAB LA PrEP when offered at public health facilities to cisgender men and transgender or gender non-binary individuals who have sex with persons assigned male at birth. The study will also evaluate two nested implementation strategies, an mHealth education and decision support tool and a WhatsApp injection appointment reminder. The study will also assess overall facilitators and barriers to integrating CAB LA into existing oral PrEP services.

DETAILED DESCRIPTION:
HIV Pre-Exposure Prophylaxis in Latin America: Results from randomized clinical trials and observational studies have proven that oral tenofovir disoproxil fumarate-based pre-exposure prophylaxis (PrEP) is protective against HIV acquisition. This protection has been confirmed to be both effective and safe across all types of exposures, sexes and gender identities, and dosing regimens. PrEP is now recommended as part of the standard prevention regimen by the World Health Organization (WHO) for individuals at substantial risk of HIV infection. Increasing PrEP access is a priority in Latin America, where several countries have recorded a rising HIV infection incidence, particularly among men who have sex with men (MSM).

In 2020, there were an estimated 930,000 people in Brazil living with HIV (PLWH). Recent studies estimate an HIV prevalence among Brazilian MSM reaching approximately 23% and rates among transgender women (TGW) surpassing 30% in some cities. Young MSM are among the few populations with increasing numbers of new HIV infections in Brazil, where HIV incidence has stabilized in overall population. PrEP in Brazil is freely available through the national Public Health System. As of May 2022, there were 424 healthcare centers across all Brazilian states providing PrEP to approximately 343,000 individuals. Although over 80% of current PrEP users in Brazil are MSM, PrEP utilization remains well below the 2018 estimate of 66,120 Brazilian MSM aged 15-64 years who were eligible for and willing to use PrEP. This number is likely to be even higher with 2021 population estimates. Among more than 57,000 individuals that initiated PrEP in Brazil, approximately 43% discontinued its use. PrEP discontinuation was common among MSM (~40%) and TGW (over 50%).

Tenofovir-based oral PrEP has been effective in dramatically reducing population-level HIV incidence in multiple districts, including London, San Francisco, New South Wales, and in rural Kenya and Ugand. Despite these successes, PrEP has not decreased HIV incidence equally, particularly among the most at-risk populations (women, youth, racial and ethnic minority MSM, and TGW), due to user adherence challenges. PrEP Brasil, the Brazilian daily oral PrEP demonstration study, identified that 74% of overall participants had protective drug levels. Nevertheless, young participants and TGW had decreasing rates of protective drug concentrations throughout the study. In addition, data from the ImPrEP study, the largest PrEP demonstration study in Latin America with the goal of evaluating the feasibility of same-day PrEP implementation to MSM and transgender women in the context of the Public Health Systems of Brazil, Mexico, and Peru, identified lower PrEP adherence among transgender woman and individuals younger than 24 years of age.

To realize PrEP benefits, individuals need to both initiate PrEP and remain on PrEP during periods at-risk. In multiple studies, reasons for stopping or never initiating PrEP include, in addition to challenges accessing the medication, low self-perceived risk, concerns about medication side effects or a desire not to take a daily pill, stigma, or competing life events. Long-acting PrEP agents have the potential to address some of these concerns by providing consistent protection through infrequent, discrete administration, avoiding relying on adherence to a daily oral regimen and the need for disclosure with sex partners and acquaintances.

Long Acting Cabotegravir for Prevention: Long-acting injectable cabotegravir (CAB-LA) is a novel integrase strand-transfer inhibitor (INSTI). Two large randomized controlled trials (RCTs), known as HIV Prevention Trials Network (HPTN) Study 083 and HPTN Study 084, have demonstrated the effectiveness of injectable cabotegravir when compared to oral tenofovir-disoproxil-fumarate/emtricitabine (TDF/FTC) PrEP.

HPTN 083 was a double-blind double-dummy RCT which assessed the effectiveness of every-8-week dosing of cabotegravir for PrEP compared to oral TDF/FTC PrEP among cisgender men and TGW at 43 sites in the United States, Latin America, Asia, and Africa using a non-inferiority study design. Overall, 4,566 participants, of whom 12.5% were TGW, were assigned 1:1 to injectable cabotegravir given every 8 weeks or daily oral TDF/FTC PrEP and were followed for 153 weeks during the blinded phase of the study. The blinded portion of the study was stopped early for efficacy, with injectable cabotegravir demonstrating statistical superiority over TDF/FTC with a hazard ratio (HR) of 0.34 for HIV incidence when compared to TDF/FTC [95% confidence interval (CI)=0.18-0.62]. Evidence of post-enrollment HIV infection was identified in 51 participants, with only 12 of the cases occurring in the cabotegravir group. When examining sub-groups, the magnitude and direction of the effectiveness of cabotegravir was preserved among populations who have historically experienced greater adherence challenges with TDF/FTC PrEP, including among youth, TGW, and U.S. Black participants.

Updated results including incident HIV infections for the Year 1 unblinded period show 11 new incident HIV infections in the CAB arm and 31 in the TDF/FTC arm, maintaining a HR of 0.34, with incidence rates in both arms showing more than 1 ½ fold higher in the unblinded period compared to the blinded period, with no new safety concerns identified. PrEP adherence declined in both arms over time. In the TDF/FTC arm, adherence decreased from 73% in the blinded period to 59% the Year 1 unblinded period. In the CAB arm, injection "coverage" declined from 91.5% during the blinded study period to 79.9% during the Year 1 unblinded period.

An important characteristic of ARV-based PrEP regimens is how long the drug persists after final administration (i.e., the tail phase of the drug). It was initially thought that the pharmacokinetic tail could create a period of vulnerability in persons who acquire HIV infection, allowing for emergence of drug-resistant strains (33,34). However, based on the current data, it seems very unlikely that this is a period of vulnerability as no incident infections have happened during the pharmacological tail period in the HTPN 083 trial.

Rare breakthrough infections were observed in HPTN 083, but detection of HIV infection in participants who received CAB PrEP was often delayed using standard HIV testing algorithms. Integrase strand transfer inhibitor (INSTI) resistance-associated mutations (RAMs) were detected in 5 CAB-exposed participants with HIV infection (GenoSure PRIME assay, viral load [VL] ≥500 c/mL); 2 other participants did not have genotyping results since all VLs were <500 c/mL. In all 7 participants, detection of infection at study sites using rapid tests and antigen/antibody tests was delayed (median 60 days; range 35-117) and all 7 participants received CAB-LA injections after HIV infection had occurred. The use of a single-genome sequencing (SGS) INSTI genotyping assay detected INSTI RAMs in 6/7 participants. The use of an RNA assay with a limit of detection (LOD) of 30 copies/mL detected infection before a major INSTI RAM was detected (4 cases) or before additional major INSTI RAMs accumulated (2 cases). In the last case, this could not be assessed since SGS was not successful before the first site-positive visit. Consistent with newly released CDC guidelines, earlier detection of HIV infection using an HIV RNA assay in the setting of CAB-LA PrEP would allow for earlier antiretroviral therapy (ART) initiation which may reduce the risk of INSTI resistance. The impact of different HIV testing strategies on INSTI resistance in real-world settings is unclear making implementation science projects critical.

Using a similar superiority study design, HPTN 084 enrolled HIV negative cisgender women at risk for HIV infection at 20 sites in 7 countries in sub-Saharan Africa including South Africa, Botswana, Eswatini, Zimbabwe, Malawi, Kenya and Uganda. Overall, 3,223 cisgender women were enrolled, with 57% of participants 18-25 years old. There were 40 confirmed HIV infections observed over 3892 person-years of follow up. The overall HIV incidence among all study participants was 1%, suggesting that both products were highly effective in preventing HIV in this population. Four infections were detected in the CAB arm which is equivalent to an incidence of 0.2%, and 36 infections were detected in participants assigned to TDF/FTC which is equivalent to an incidence of 1.85%. No differences in treatment effects were observed in pre-specified sub-group analyses exploring effects by age, BMI, and contraceptive use.

Data from 083 and 084 supported the US Food and Drug Administration regulatory approval of CAB-LA for HIV prevention on December 20, 2021. Subsequently, national regulatory approval for CAB-LA PrEP has been sought in numerous countries, including Brazil.

The ImPrEP Study: ImPrEP is a UNITAID funded, multi-country PrEP implementation project. It is a collaboration between the Oswaldo Cruz Foundation (Fiocruz) and Ministries of Health from Brazil, Peru, and Mexico. One of the ImPrEP components has been a multi-site prospective, open-label demonstration study to assess uptake, acceptability, and feasibility of same-day, daily TDF/FTC oral PrEP among MSM and TGW at substantial risk for HIV acquisition. A total of 28 sites conducted the study, 14 sites in Brazil, 4 in Mexico, and 10 in Peru. Overall, a total of 9,509 participants were enrolled with 26% being young (18-24 years), 73% were non-white, and over 640 (5.6%) participants were TGW. Overall, 68% of participants had long-term engagement; however, younger, less educated participants, TGW and sex workers were significantly less likely to reach long-term engagement.

Although HIV incidence during the study was relatively low (0.82/100 person-years), it was higher among non-white, younger (18-24 years) and TGW participants. These disproportionately worse outcomes highlight that PrEP agents not requiring daily or planned oral dosing could increase effective PrEP use among these most vulnerable populations. It is reassuring that injectable cabotegravir has demonstrated comparable effectiveness among youth, Black MSM, and TGW in clinical trials. However, advantages in bypassing daily adherence behavior may not be realized if individuals cannot access injectable PrEP or do not return for repeat injections. Additional data from injectable PrEP service delivery in real-world settings will be needed to support roll-out and national program decisions to include CAB LA PrEP as part of prevention services.

Person-centered HIV Prevention: At the core of person-centered HIV prevention is the acknowledgement that people are best placed to decide which prevention methods are right for them and that their preference may change over the course of their life. Person-centered care emphasizes meeting an individual's sexual preferences, needs, and goals, using person-centered counseling approaches, such as shared decision-making. In a counseling visit utilizing shared decision-making, the individual is recognized as the expert regarding their lived experience, life situations, needs, and preferences for sexual health prevention and care. The conclusion of such a counseling conversation may include patients choosing not to use a prevention method or discontinuation of a more effective method for a less effective method (or no method at all). Central to a people-centered approach to HIV prevention is effectively communicating information about the advantages and disadvantages of available methods and about product characteristics to facilitate informed decision making. A people-centered approach also supports adherence, once an HIV prevention method has been chosen, in ways which will be experienced as supportive and useful by the method user.

Implementation Research is Needed to Prepare for Scale-up of CAB-LA PrEP: Now that the efficacy of CAB-LA PrEP has been proven in large clinical trials, implementation studies must explore how to best integrate its delivery into existing PrEP services in 'real world' settings. Implementation studies provide crucial information about how interventions, proven efficacious under randomized clinical trial conditions, can be optimized for delivery within routine service contexts. Implementation research provides an opportunity to identify implementation barriers and to maximize the feasibility and acceptability of intervention delivery as well as intervention effectiveness.

The investigators are proposing a CAB-LA implementation-effectiveness research study (hybrid Type 2) that leverages the impact of the current ImPrEP project in Brazil to generate critical evidence about the feasibility, acceptability, and effectiveness of incorporating CAB-LA PrEP into existing services for oral PrEP. This implementation project is fully grounded in the principles of people-centered care, with a focus on respect for participant's preference and expressed needs. Study results will inform global guideline recommendations, regional and national policy development, and program implementation guidance for Brazil and other low and middle-income countries (LMIC).

In the field of contraception, increased availability of method options and informed decision-making about method choice has improved uptake and persistence of the contraceptive methods used. It is likely that expanding method options for HIV prevention will similarly improve uptake and persistence. However, informed decision-making requires user understanding of how methods must be used, potential side effects, and effectiveness. Although health worker counseling plays a crucial role in providing patients with information about different methods, mobile health (mHealth) has great potential to provide valuable additional educational support. For example, decision support tools have been shown to be both acceptable and effective in guiding women's contraceptive decisions. The investigators will develop and test a similar mHealth education and decision support tool for use in MSM, non-binary and transgender populations.

Adherence to the CAB LA injection schedule (at 1 month for a second dose, and every 2 months thereafter) will be crucial to preventing HIV acquisition. Although the results of HPTN 083 and 084 demonstrated that overall, participants had better adherence to clinic visits for their CAB LA injections than for daily oral PrEP, additional support for maintaining adherence to the CAB LA injection clinic visits is needed for some users. In a randomized controlled trial, interactive short message service (SMS)-based support improved daily oral PrEP persistence (80% vs. 57% at 36 weeks, p<0.01) when compared to standard of care among diverse young MSM at risk for HIV acquisition in the US. In the current study, The investigators will test the impact of WhatsApp appointment reminders on participant adherence and continuation of CAB-LA PrEP.

Finally, this implementation research study will include an exploration of the best, acceptable HIV testing strategy and algorithm for use with CAB LA PrEP. A key challenge with the implementation of injectable cabotegravir as PrEP is its impact on diagnosis of breakthrough HIV infections. Detection of HIV infection at study sites was delayed in participants in both HPTN 083 and 084, illustrating the challenge of using conventional testing approaches to screen for HIV infection in studies using potent, long-acting PrEP agents. With CAB-LA, the result of delayed diagnosis may contribute to the development of resistance associated mutations that would be expected to confer reduced susceptibility to integrase inhibitors. The use of an HIV RNA assay for screening could possibly detect these infections earlier, prompting earlier ART initiation and preventing emergence of HIV resistance. Nevertheless, viral load (VL) testing is expensive and could cause implementation of cabotegravir-based PrEP to remain limited in LMICs should these testing requirements be adopted by regulatory agencies and guideline panels. Early detection of HIV infection and prompt ART initiation could improve clinical outcomes in persons who become infected despite CAB-LA prophylaxis. In addition to HIV rapid tests this study will incorporate the use of point-of-care VL testing with GeneXpert for VL to identify HIV infection not detectable with the HIV rapid tests at enrollment. The use of this technology will enable participants to receive VL results and, if negative, receive a same-day CAB LA injection. The use of non-INSTI ART to treat people who acquire HIV while taking injectable CAB may be an option.

ELIGIBILITY:
Inclusion Criteria:

1. Cisgender men, non-binary (assigned as male at birth) or transgender women and men
2. Report having anal sex with a person assigned male at birth in the last six months (Persons born female having sex only with other persons born female are excluded)
3. Age 18-30 years
4. Seek a study clinic looking for PrEP
5. CAB LA and TDF/FTC PrEP naïve
6. Willing and able to provide written informed consent and adhere to the study requirements
7. Non-reactive / negative HIV test results, including both HIV rapid tests and an undetectable HIV RNA at enrollment for individuals choosing injectable CAB-LA.
8. No report of hepatic dysfunction. Candidates reporting liver disease will have their enrollment visit postponed until laboratory results of liver function are available. Individuals with ALT >=5x ULN, OR ALT>=3xULN and bilirubin >=1.5xULN will be excluded. See section 7 (Study Procedures - Enrollment visit).
9. Willing to undergo all required study procedures.

Exclusion Criteria:

1. One or more reactive or positive HIV test result at enrollment visit, even if HIV infection is not confirmed.
2. Currently participating in interventional trial of PrEP agents, HIV vaccine trial or experimental medication.
3. Positive pregnancy test, breastfeeding, or intention to become pregnant at enrolment (for transgender men).
4. Prior participation in studies with Cabotegravir.
5. A history or presence of allergy to the study drug components.
6. Past participation in HIV vaccine trial. An exception will be made for participants that can provide documentation of receipt of placebo (not active arm).
7. Plan to relocate out of the area during the study period.
8. Surgically placed or injected buttock implants or fillers, per self-report.
9. Has a dermatological/inflammatory skin condition overlying the buttock region which in the opinion of the study investigator, in consultation with the Clinical Study Coordination (CSC), may interfere with interpretation of injection site reactions.
10. Active or planned use of contraindicated co-administered for which significant decreases in Cabotegravir plasma concentrations may occur due uridine diphosphate glucuronosyltransferase (UGT1A1):

    * Anticonvulsants: Carbamazepine, Oxcarbazepine, Phenobarbital, Phenytoin
    * Antimycobacterials: Rifampin, Rifapentine *Any prohibited medications that decrease CAB concentrations should be discontinued for a minimum of four weeks or a minimum of three half-lives (whichever is longer) prior to the first dose.
11. Current or anticipated need for chronic systemic anticoagulation or a history of known or suspected bleeding disorder, including a history of prolonged bleeding.
12. History of severe hepatic impairment (including but not limited to a history of liver failure or hospitalization for liver disease, a history of hepatocellular carcinoma or near liver transplant).
13. Individuals with advanced Hepatitis C.
14. Other medical conditions that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men, non-binary (assigned as male at birth) or transgender women and men
Enrollment: 1200 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incident HIV infection | 2 years
  Among individuals who test positive on HIV rapid test, midpoint between last negative HIV rapid test and first HIV positive rapid test

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Grinsztejn, MD, PhD, Principal Investigator — Instituto Nacional de Infectologia Evandro Chagas/ FIOCRUZ; Valdilea Veloso, MD, PhD, Study Director — Instituto Nacional de Infectologia Evandro Chagas/ FIOCRUZ
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas/ FIOCRUZ, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Pimenta C, Mann CG, Hoagland B, Carvalheira E, Jalil C, Benedetti M, Fernandes N, Coutinho C, Jalil EM, Secco Torres Silva M, Trefiglio R, Farias A, Mourao MPG, Madruga JV, de Lima JN, Zonta R, O'Malley G, Veloso VG, Grinsztejn B, Torres TS; ImPrEP CAB-Brasil Study. Exploring perceptions and preferences for PrEP choice and of an mHealth intervention: insights from the ImPrEP CAB-Brasil study. J Int AIDS Soc. 2025 Jul;28 Suppl 2(Suppl 2):e26493. doi: 10.1002/jia2.26493. PMID 40600468
- [Derived] Grinsztejn B, Torres TS, Hoagland B, Jalil EM, Moreira RI, O'Malley G, Shade SB, Benedetti MR, Moreira J, Simpson K, Pimenta MC, Veloso VG; ImPrEP CAB-Brasil Study Team. Long-Acting Injectable Cabotegravir for HIV Preexposure Prophylaxis Among Sexual and Gender Minorities: Protocol for an Implementation Study. JMIR Public Health Surveill. 2023 Apr 19;9:e44961. doi: 10.2196/44961. PMID 37074775
- See also: WHO. Consolidated guidelines on the use of antiretroviral drugs for treating and preventing HIV infection. Second Edition. Recommendations for a public health approach — https://www.who.int/hiv/pub/arv/arv-2016/en/
- See also: UNAIDS. New HIV infections rising in Latin America-key populations particularly affected [Internet]. 2019 [cited 2022 Apr 21]. — https://www.unaids.org/en/resources/presscentre/featurestories/2019/october/20191014_latin-america
- See also: UNAIDS. Global Aids Strategy 2021 - 2026 End Inequalities . End Aids . Unaids [Internet]. 2021;160 — https://www.unaids.org/en/Global-AIDS-Strategy-2021-2026
- See also: United Nations Programme on HIV/aids. UNAIDS. UNAIDS data 2021. 2021;4-38. — https://www.unaids.org/sites/default/files/media_asset/JC3032_AIDS_Data_book_2021_En.pdf